CLINICAL TRIAL: NCT04483674
Title: Bictegravir/FTC/TAF for the Treatment of Primary HIV Infection
Acronym: BIC-PHI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anna Cruceta (Other)
Responsible Party: Sponsor-Investigator, Anna Cruceta, Project Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-000601-89
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: HIV Primary Infection
Keywords: Human Immunodeficiency Virus; HIV Primary Infection; Biktarvy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — bictegravir; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biktarvy (Experimental): Patients will receive one pill with 50mg bictegravir/200mg emtricitabine /25mg tenofovir alafenamide orally once a day, for 48 weeks
  Interventions: Drug: 50mg bictegravir/200mg emtricitabine/25mg tenofovir alafenamide

INTERVENTIONS:
Drug: 50mg bictegravir/200mg emtricitabine/25mg tenofovir alafenamide — Patients will be administered one pill of 50mg bictegravir/200mg emtricitabine/25mg tenofovir alafenamide daily for 48 weeks with regular check-ups at weeks 4,8,12,24 and 48 including:
  * complete physical examination
  * register concomitant medication
  * blood test
  * concomitant medications
  * assessment od adverse events
  * assessement of compliance
  * PSQI and CESTA questionnaire (week 4 and 48)
  * Recommendation in contraception methods
  * Stool sample and pregnancy test urine (week 0 and 48)
  The total of blood required for each visit is 30ml except the visit of week 48 (90ml) The total of urine required is 6 mL
  Other Names: Biktarvy

SUMMARY:
The purpose of this study is to assess the efficacy of Bictegravir/FTC/TAF in patients with less of 100 days post HIV infection

DETAILED DESCRIPTION:
After providing informed consent, patients will undergo to a screening visit. If they meet the inclusion criteria and none of the exclusion will be included in this trial. Patients will take one tablet of Biktarvy at day for 48 weeks. Then the results will be compared with a cohort of 66 patients treated with 2 nucleoside analogues and one integrase chain transfer inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-65 years
* ART naïve
* HIV infection of less than 100 days post-infection (documented 3 month previous negative serology or incomplete WB test with negative p31 band)
* Women of child-bearing potential must have a negative pregnancy test in serum before the inclusion in the study and agree to use highly effective contraceptive methods, including intrauterine device, bilateral tubal occlusion or a vasectomized partner.

Exclusion Criteria:

* Known hypersensitivity to any drug included in Bictegravir/FTC/TAF regimen
* AST >5 times UNL
* Creatinine Clearance <30 mL/min/1.73m2
* Any end-stage organ disease
* Acute or chronic HCV co-infection
* Use of PrEP with Truvada® until 4 weeks before the onset of symptoms of PHI (risk of acquired-drug resistance to FCT or TDF).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Portion of patients with a VL (viral load)< 50 Copies at week 48 | 48 weeks
  Portion of patients with rapid ART (Antiretroviral therapy) initiation who reached a VL< 50 copies at 48 week in the intention to treat population determined by PCR

SECONDARY OUTCOMES:
Viral Load at 4,8,12,24 y 48 weeks | weeks 4,8,12,24,48
  Determination by PCR (Polymerase Chain Reaction) of viral load at differents weeks of treatment
Portion of patients with > 900 cells CD4+ | weeks 24 and 48
  Proportion of patients with >900 cells CD4+
Days elapsed between diagnosis and bictegravir/FTC/TAF initiation | week 48
  Days elapsed between diagnosis and bictegravir/FTC/TAF initiation, day elapsed between first clinical visit and Bictegravir/FTC/TAF initiation
Proportion of patients treated with Bictegravir/FTC/TAF who reached a VL<50 copies at 48 weeks in the intention-to-treat (ITT) population | week 48
  Proportion of patients treated with Bictegravir/FTC/TAF who reached a VL<50 copies at 48 weeks in the intention-to-treat (ITT) population in comparison with other InSTI-, based ART regimens
AE (adverse event) leading to discontinuation rate | week 48
  AE leading to discontinuation rate in comparison with other InSTI- based ATR regimens
CD4, CD4/CD8 ratio | weeks 4,8,12,24,48
  CD4, CD4/CD8 ratio at weeks 4,8,12,24 and 48
AE rate | week 48
  AE rate (overall and AE leading to discontinuation)
Number of required regimen changes | week 48
  Number of required regimen changes stratified by: adverse events/toxicity, virological failure, simplification, transmitted drug resistance (including polymorphisms for InSTIs).
Quality of life and satisfaction: questionnaire | day 0, week 4 and 48
  Quality of life and satisfaction evaluated through a CESTA questionnaire (Spanish Questionnaire of Satisfaction whit Antiretroviral Treatment) at 4 and 48 weeks (or at the end of study in case of early termination) of the study period, and Pittsburgh Sleep Quality Index (PSQI) at day 0, 4 week and 48 weeks (or at the end of study in case of early termination) of the study period
Viral reservoir, inflammatory and immunological markers and fecal microbiome composition | weeks 0,48
  Viral reservoir, inflammatory and immunological markers and fecal microbiome composition

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain